CLINICAL TRIAL: NCT05248360
Title: A Randomized, Double-blind, Crossover, Placebo-controlled Study to Evaluate the Efficacy and Safety of Hydrogen-oxygen Mixed Gas in the Treatment of Insomnia
Brief Title: Hydrogen-oxygen Mixed Gas in the Treatment of Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chun-Feng Liu, Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JD-LK-2021-100-03
Record Dates: First submitted 2022-02-03; First posted 2022-02-21 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Insomnia
Keywords: Insomnia; Hydrogen-oxygen Mixed Gas
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Hydrogen-oxygen mixed gas(H2-O2, 66.6% hydrogen, 33.3% oxygen) inhalation, 900ml/min, 2h/d
  Interventions: Device: Hydrogen-oxygen mixed gas(H2-O2) inhalation
- Control group (Placebo Comparator): Air inhalation, 900ml/min, 2h/d
  Interventions: Device: Air inhalation

INTERVENTIONS:
Device: Hydrogen-oxygen mixed gas(H2-O2) inhalation — H2-O2 inhalation, 900ml/min, 2h/d * 4 weeks (≥5 days/week)
  Arms: Experimental group
Device: Air inhalation — Air inhalation, 900ml/min, 2h/d * 4 weeks (≥5 days/week)
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hydrogen-oxygen mixed gas inhalation in the treatment of insomnia.

DETAILED DESCRIPTION:
This ia a randomized, double-blind, crossover, placebo-controlled Study. The purpose is to evaluate the efficacy and safety of hydrogen-oxygen mixed gas(H2-O2) inhalation in the treatment of insomnia, and explore the possible mechanism by detecting the changes of serum inflammatory factors (CRP, IL-6, IL-1β, TNF-α) levels, so as to seek an effective therapy for insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of insomnia according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
2. No use of sleep medications within the preceding 2 weeks, or a stable dose of only one sedative hypnotic medicine for at least 1 month before the enrollment and remain unchanged throughout the course of the study.
3. Signed informed consent form (ICF).

Exclusion Criteria:

1. Complicated with other sleep disorders (sleep apnea syndrome, narcolepsy, restless legs syndrome, nocturia, etc.);
2. Complicated with serious heart, lung, liver or renal diseases or malignant tumor;
3. History of mental illness;
4. Drugs or substances abuse;
5. Pregnant women, breast-feeding women or those with recent birth plans;
6. Participants in other clinical trials within 1 month before the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in sleep efficiency by polysomnography (PSG) at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' sleep quality.
Change from baseline in total sleep time by PSG at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' sleep quality.
Change from baseline in sleep latency by PSG at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' sleep quality.
Change from baseline in wake time after sleep onset by PSG at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' sleep quality.
Change from baseline in Insomnia Severity Index (ISI) score at 14 weeks | visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The ISI is widely used to measure the severity of Insomnia. The ISI score ranges from 0 to 28. The higher the ISI score is, the worse the symptoms are.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) score at 14 weeks | visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The PSQI is widely used to measure sleep quality. The PSQI score ranges from 0 to 21. The higher the PSQI score is, the worse the sleep quality is.

SECONDARY OUTCOMES:
Change from baseline in Hamilton Anxiety Scale (HAMA) score at 14 weeks | Visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The HAMA is a widely used interview scale to measure the severity of anxiety. The HAMA score ranges from 0 to 56. The higher the HAMA score is, the worse the symptoms are.
Change from baseline in Hamilton Depression Scale-17 (HAMD-17) score at 14 weeks | Visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The HAMD-17 is a test measuring the severity of depressive symptoms. The HAMA-17 score ranges from 0 to 52. The higher the HAMA score is, the worse the symptoms are.
Change from baseline in Mini-Mental State Examination (MMSE) score at 14 weeks | Visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The MMSE is widely used to assess cognition. The MMSE score ranges from 0 to 30. The higher the HAMA score is, the better the cognitive function is.
Change from baseline in Montreal Cognitive Assessment (MOCA) score at 14 weeks | Visit 1(baseline), visit 3(4th week), visit 4(6th week), visit 6(10th week), visit 7(14th week)
  The MoCA is widely used to assess cognition. The HAMA-17 score ranges from 0 to 30. The higher the HAMA score is, the better the cognitive function is.
Change from baseline in C-reactive protein (CRP) at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' serum inflammatory factor.
Change from baseline in Interleukin-6 (IL-6) at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' serum inflammatory factor.
Change from baseline in Interleukin-1β ( IL-1β) at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' serum inflammatory factor.
Change from baseline in tumor necrosis factor-α (TNF-α) at 10 weeks | visit 1(baseline), visit 3(4th week), visit 6(10th week)
  This outcome reflects change of patients' serum inflammatory factor.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, MD, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin MR, Olmstead R, Carroll JE. Sleep Disturbance, Sleep Duration, and Inflammation: A Systematic Review and Meta-Analysis of Cohort Studies and Experimental Sleep Deprivation. Biol Psychiatry. 2016 Jul 1;80(1):40-52. doi: 10.1016/j.biopsych.2015.05.014. Epub 2015 Jun 1. PMID 26140821
- [Background] Ohta S. Molecular hydrogen as a novel antioxidant: overview of the advantages of hydrogen for medical applications. Methods Enzymol. 2015;555:289-317. doi: 10.1016/bs.mie.2014.11.038. Epub 2015 Jan 21. PMID 25747486